CLINICAL TRIAL: NCT07107542
Title: Entrustable Professional Activities and Mini-Clinical Evaluation Exercise in a Simulated Workplace-based Assessment for Physical Occupational Therapist Intern
Brief Title: Exploring the Relationship Between Mini-Clinical Evaluation Exercise (Mini-CEX) and Entrustable Professional Activities (EPAs) in Occupational Therapy Clinical Interns' Independent Competence
Status: Not yet recruiting | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chao-Yi Cheng, Occupational Therapist, Department of Rehabilitation, Far Eastern Memorial Hospital, Far Eastern Memorial Hospital
Other Study IDs: 114026-E
Record Dates: First submitted 2025-07-11; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Entrustable Professional Activities; Mini-clinical Evaluation Exercise; Physical Occupational Therapy; Occupational Therapy Education
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Occupational Therapy Fieldwork Interns: This group includes occupational therapy interns specializing in the physical domain who are undergoing fieldwork training at Far Eastern Memorial Hospital. Participants are recruited during their sixth week of internship and assessed at the eighth week. The study evaluates their fieldwork performance using Mini-Clinical Evaluation Exercise (Mini-CEX) and Entrustable Professional Activities (EPAs) as standard assessment tools. Participation is voluntary with informed consent, and no additional interventions beyond routine fieldwork training are applied. Data collected will be used to analyze the relationship between these assessment tools and interns' readiness for independent practice.
  Interventions: Other: Mini-Clinical Evaluation Exercise (Mini-CEX) and Entrustable Professional Activities (EPAs) Assessment

INTERVENTIONS:
Other: Mini-Clinical Evaluation Exercise (Mini-CEX) and Entrustable Professional Activities (EPAs) Assessment — Participants undergo standard fieldwork assessments using Mini-CEX and EPAs during their internship to evaluate fieldwork competence and readiness for independent practice. These are observational assessments without additional experimental interventions.

SUMMARY:
The goal of this observational cross-sectional study is to evaluate whether the combined use of Mini-Clinical Evaluation Exercise (Mini-CEX) and Entrustable Professional Activities (EPAs) can assess the independent clinical competence of occupational therapy interns at Far Eastern Memorial Hospital. The main questions it aims to answer are:

1. Does the performance on Mini-CEX correlate with the interns' ability to perform independently?
2. Does the use of EPAs provide additional insight into interns' readiness for unsupervised clinical practice?

Participants will:

1. Provide informed consent at the sixth week of their internship.
2. Undergo assessment with Mini-CEX and EPAs during their eighth week of clinical training.
3. Complete demographic questionnaires including age, gender, study habits, prior university experience, parental occupation, and residence area.

DETAILED DESCRIPTION:
Medical graduates in the healthcare field apply theoretical knowledge gained during their education combined with clinical supervision to develop professional skills necessary for patient care. To comprehensively evaluate interns' professional competence during clinical training, workplace assessment tools such as the Mini-Clinical Evaluation Exercise (Mini-CEX) are commonly used. Mini-CEX, developed by the American Medical Association, assesses seven core clinical skills over a 20 to 30-minute observation period. However, Mini-CEX alone may not fully capture the interns' ability to perform independently.

Competency-Based Medical Education (CBME) emphasizes the development of core competencies, and Entrustable Professional Activities (EPAs) have been proposed as a framework to describe tasks that trainees should be entrusted to perform unsupervised at various training stages. EPAs assess the level of supervision required, reflecting the degree of trust clinical supervisors place in trainees. In Taiwan, EPAs tailored for occupational therapy have been developed and implemented under the guidance of the Occupational Therapy Association.

This study aims to explore the relationship between Mini-CEX and EPAs in evaluating occupational therapy interns' independent clinical competence. The study will recruit 50 interns from the physiological domain of occupational therapy at Far Eastern Memorial Hospital over four years. Participants will be recruited at the sixth week of their internship, provide informed consent, and be assessed at the eighth week using both Mini-CEX and EPAs. The assessments are part of routine clinical training evaluations and take approximately 20 minutes.

Data collected will include demographic information and assessment scores. Statistical analyses will involve descriptive statistics, Pearson correlation to examine relationships between variables, and multiple linear regression to identify predictors of clinical performance, including age, gender, study habits, prior university experience, parental occupation, and residence area. Participation is voluntary and will not affect interns' clinical training or evaluation outcomes.

This study seeks to provide evidence on whether combining Mini-CEX and EPAs offers a more reliable assessment of interns' readiness for independent clinical practice, potentially informing future educational strategies in occupational therapy training.

ELIGIBILITY:
Inclusion Criteria:

* Occupational therapy interns in the physical domain at Far Eastern Memorial Hospital
* Provide informed consent to participate

Exclusion Criteria:

* None specified

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study population consists of occupational therapy interns undergoing physical domain fieldwork at Far Eastern Memorial Hospital. Participants are typically fourth-year students engaged in clinical internship training.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-08 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Independent Clinical Competence of Occupational Therapy Interns | Assessment conducted at the eighth week of internship fieldwork.
  The primary outcome is the assessment of occupational therapy interns' independent performance during fieldwork, measured by combined scores of the Mini-Clinical Evaluation Exercise (Mini-CEX) and Entrustable Professional Activities (EPAs). The Mini-CEX evaluates seven core clinical competencies, scored from 1 to 9 per item, with higher scores indicating better clinical performance. EPAs assess competence based on supervision levels, scored from 1 to 5, where higher scores reflect greater independence and readiness for unsupervised clinical practice. This combined assessment captures interns' clinical skills, decision-making, and preparedness for independent work.

SECONDARY OUTCOMES:
Correlation of Demographic Factors with fieldwork Competence | Data collected and analyzed at the eighth week of internship.
  Analysis of demographic variables including age, gender, average study time, prior university experience, parental occupation, and residence area, to explore their association with interns' performance on Mini-CEX and EPAs assessments.

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
This study will not share individual participant data (IPD) due to considerations related to participant privacy and confidentiality. The data collected involve sensitive personal and demographic information of occupational therapy interns, and sharing such data could risk identification despite de-identification efforts. Additionally, the study was conducted under ethical approvals that restrict data sharing beyond the research team. Aggregate results and summary findings will be made publicly available through publications and ClinicalTrials.gov, ensuring transparency while protecting participant rights.

REFERENCES:
- [Background] Ten Cate O, Chen HC, Hoff RG, Peters H, Bok H, van der Schaaf M. Curriculum development for the workplace using Entrustable Professional Activities (EPAs): AMEE Guide No. 99. Med Teach. 2015;37(11):983-1002. doi: 10.3109/0142159X.2015.1060308. Epub 2015 Jul 14. PMID 26172347
- [Background] Pinilla S, Kyrou A, Kloppel S, Strik W, Nissen C, Huwendiek S. Workplace-based assessments of entrustable professional activities in a psychiatry core clerkship: an observational study. BMC Med Educ. 2021 Apr 21;21(1):223. doi: 10.1186/s12909-021-02637-4. PMID 33882926
- [Background] Fu, C. P., Chiang, F. M., Lee, C. Y., Chi, H. Y., Wu, J. L., Lin, Y. J., Li, M. W., Chen, Y. J., Chang, W. Y., Chang, W. D., Huang, S. M., Liao, W. S., Yang, Y. C., Huang, C. K., Kuo, N. J., Liu, T. H., & Chen, Y. L. (2023). Developing the topics of entrustable professional activities in pediatric occupational therapy in Taiwan: A pilot study. Taiwan Journal of Occupational Therapy, 41(2), 91-110. https://doi.org/10.6594/tjot.202308_41(2).0001
- See also: Official website of the rehabilitation research team. This site does not currently contain detailed information about this specific study. For study-related inquiries, please contact the research team directly. — https://sites.google.com/view/femhrehab/%E6%9C%AC%E7%A7%91%E4%BB%8B%E7%B4%B9/%E9%86%AB%E7%99%82%E5%9C%98%E9%9A%8A%E4%BB%8B%E7%B4%B9
- Available data/document: Study Protocol — https://sites.google.com/view/femhrehab/%E6%9C%AC%E7%A7%91%E4%BB%8B%E7%B4%B9/%E9%86%AB%E7%99%82%E5%9C%98%E9%9A%8A%E4%BB%8B%E7%B4%B9 — This document contains the study protocol and statistical analysis plan for the cross-sectional study assessing Mini-CEX and EPAs in occupational therapy interns.

DOCUMENTS (2):
  • Study Protocol (2025-03-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT07107542/Prot_000.pdf
  • Informed Consent Form (2025-03-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT07107542/ICF_001.pdf